CLINICAL TRIAL: NCT04759716
Title: The Effectiveness of Health Literacy-based Weight Control Intervention Via Mobile Health Application for Overweight and Obese Adolescent: A Longitudinal Panel Study
Brief Title: Health Literacy-based Weight Control Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201912048RIND
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Overweight
Keywords: weight control; Adolescents; overweight; obesity; Mobile health
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Literacy-based Weight Control Intervention arm (Experimental): intervention arm will receive weight control program
  Interventions: Other: Health Literacy-based Weight Control Intervention
- control arm (No Intervention): routine care

INTERVENTIONS:
Other: Health Literacy-based Weight Control Intervention — intervention arm will be applied to receive health literacy-based mobile Health App, smart sports watch Fitbit versa during the 12 months weight control program
  Arms: Health Literacy-based Weight Control Intervention arm

SUMMARY:
This research will be a continuation of 2015-2017 research projects of smart phone APP research granted by Ministry of Science and Technology. First of all, a four-wave-cross-sectional survey by cluster sampling is used to recruit 90 adolescents aged 13-19 from high school, vocational schools or colleges to test the feasibility of the health literacy-based weight-control program. In the second stage, a two-arm randomized controlled trial (RCT) will be applied to recruit 240 overweight or obese teenagers to receive health literacy-based mobile Health App, smart sports watch Fitbit versa during the 12 months weight control program. Based on the previous research evidences, the outcome follow up will be scheduled on 3 months, 9 months, 15 months, and 21 months after the mobile Health Apps intervention. Short-term outcome indicators include health literacy, diet pattern, and dietary behaviors; long-term outcome indicators include BMI z-score, waist circumference. Intention-to-treat analysis, generalized linear mixed models with repeated measures, multiple regression analysis model, and counterfactual causal Inference will be applied to analyze the effectiveness of the interventions.

DETAILED DESCRIPTION:
Adolescent overweight and obesity are major health issues and challenges worldwide. According to the estimate of World Health Organization, the number of obese people in the world has tripled since 1975. Overweight and obese children and adolescents increased from 124 million in 1975 to 340 million in 2016. The obese young children will have a negative impact on the physical, psychological and social health, and will increase the risk of obesity in adulthood.

This study is a continuing project of the research funded by the Ministry of Science and Technology to explore the smartphone app, health literacy. Purposes of this study are to (1) validate the Health literacy based mobile Health Apps Interventions, (2) conduct the mobile health apps and smart sports watches to intervene in 12 months and evaluate the effectiveness by follow-up repeated measures.

Eligibility criteria. The inclusion criteria are 13-19 years old adolescents; Could use their mobile phones to upload diet records and photos; and Adolescents and their parents agree to involve in the study and sign the consent form.

Exclusion conditions are the adolescent who with severe diseases (such as tumors and other diseases); and they already participate in other weight control program.

Methods This research will be a continuation of 2015-2017 research projects of smart phone APP research granted by Ministry of Science and Technology. First of all, a four-wave-cross-sectional survey by cluster sampling is used to recruit 90 adolescents aged 13-19 from high school, vocational schools or colleges to test the feasibility of the health literacy-based weight-control program. In the second stage, a two-arm randomized controlled trial (RCT) will be applied to recruit 240 overweight or obese teenagers to receive health literacy-based mobile Health App, smart sports watch Fitbit versa during the 12 months weight control program. Based on the previous research evidences, the outcome follow up will be scheduled on 3 months, 9 months, 15 months, and 21 months after the mobile Health Apps intervention. Short-term outcome indicators include health literacy, diet pattern, and dietary behaviors; long-term outcome indicators include BMI z-score, waist circumference. Intention-to-treat analysis, generalized linear mixed models with repeated measures, multiple regression analysis model, and counterfactual causal Inference will be applied to analyze the effectiveness of the interventions.

Expected outcomes This study applies health literacy-based mobile Health Apps weight control program for the overweight and obese adolescents. By strengthening healthy lifestyle of healthy dietary pattern and physical activity for adolescents, we hope to effectively prevent adolescent obesity, so as to reduce the impacts of obesity to social, medical and economic burdens.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years old adolescents;
* Could use their mobile phones to upload diet records and photos;
* Adolescents and their parents or legal representatives agree to involve in the study and sign the consent.

Exclusion Criteria:

* Severe diseases;
* Participate in other weight control program.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
BMI(body mass index) | Change from baseline body mass index at 3 months, 9 months, 15 months, and 21 months.
  BMI = weight / height².

SECONDARY OUTCOMES:
WHR(waist-to-hip ratio ) | Change from baseline waist-to-hip ratio at 3 months, 9 months, 15 months, and 21 months.
  waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement ( W⁄H).

CONTACTS AND LOCATIONS:
Overall Officials: Bih-Shya Gau, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YH, Tzeng YF, Gau BS. Mobile Health-Based Health Literacy Weight Management Intervention Using Smart Devices for Adolescents: A Convergent Mixed-Methods Pilot Study. Nurs Health Sci. 2024 Dec;26(4):e13172. doi: 10.1111/nhs.13172. PMID 39428322